CLINICAL TRIAL: NCT05998837
Title: Single-center, Randomized, Controlled Study to Evaluate the Effects of a Six-month Treatment With Renal Glucose Transport Inhibitor (SGLT2i) Drugs on Markers of Senescence, Inflammation and Tubulointerstitial Damage in the Kidney of Patients With Chronic Kidney Disease With or Without Type 2 Diabetes
Brief Title: GLUcose Transport and REnalPROtection in Chronic Kidney Disease
Acronym: GLUTREPRO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Francesca Viazzi, Professor, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D169AL00005
Record Dates: First submitted 2023-04-16; First posted 2023-08-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease; Diabetes Mellitus, Type 2; Hypertension
Keywords: gliflozine; senescence; BOLD MRI; Blood pressure variability
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Hypertension | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Allocation to treatment group will be done by stratified randomization for diabetics and non-diabetics.
  The randomization list will be generated with a designed computer program.
Who Masked: Participant, Investigator
Masking Description: Once eligibility is verified, the Investigator will randomize the subject contacting by e-mail the Secretarial Office of the Nephrologic Clinic of the Ospedale Policlinico San Martino The assigned randomization number will communicated via e-mail and recorded by the Investigator in the CRF. Therefore both investigators and participants will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Type 2 Diabetes Dapagliflozin 10 mg (Active Comparator): Patients with Type 2 Diabetes allocated to Dapagliflozin 10 mg
  Interventions: Drug: Dapagliflozin 10mg Tab
- Type 2 Diabetes Placebo (Placebo Comparator): Patients with Type 2 Diabetes allocated to Placebo
  Interventions: Drug: Placebo
- Without Diabetes Dapagliflozin 10 mg (Active Comparator): Patients without Type 2 Diabetes allocated to Dapagliflozin 10 mg
  Interventions: Drug: Dapagliflozin 10mg Tab
- Without Diabetes Placebo (Placebo Comparator): Patients without Type 2 Diabetes allocated to Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin will be add on RAAS-i titrated with the aim to reach optimal blood pressure control as defined by European Society of Hypertension (i.e., 120-130/70-80 mmHg) in all subject.
  Prior to randomization all the patient with Type 2 Diabetes must have undergone at least 4 weeks of therapy with metformin and/or repaglinide
  Arms: Type 2 Diabetes Dapagliflozin 10 mg; Without Diabetes Dapagliflozin 10 mg
Drug: Placebo — Placebo will be add on RAAS-i titrated with the aim to reach optimal blood pressure control as defined by European Society of Hypertension (i.e., 120-130/70-80 mmHg) in all subject.
  Prior to randomization all the patient with Type 2 Diabetes must have undergone at least 4 weeks of therapy with metformin and/or repaglinide
  Arms: Type 2 Diabetes Placebo; Without Diabetes Placebo

SUMMARY:
This is a single-center, double blind, randomized, parallel-arms study designed to investigate the effects of a six-month treatment with the SGLT2i dapagliflozin on markers of kidney senescence, inflammation and tubulointerstitial damage compared to placebo. These mechanisms of renal damage will be investigated in proximal tubular epithelial cells (PTECs) isolated from urine from patients with CKD with or without T2DM and in renal biopsy specimens in a subgroup of patients with diabetic kidney disease.

DETAILED DESCRIPTION:
In the run-in phase, clinical parameters will be optimized by the use of metformin/repaglinide and or RAAS-I on the basis of the presence/absence of a diagnosis of diabetes. Subsequently, patients will be randomly assigned to start with standard therapy and placebo or dapagliflozin at the dose of 10 mg and will continue the assigned treatment for 24 weeks in double-blind and with dapagliflozin at the dose of 10 mg for an additional 48 weeks in open-label/Extended treatment.

Urine samples will be collected at T0, T1, T2, T3 and T4 and used as a source of PTECs in order to study the expression of mediators of senescence, fibrosis and inflammation in the kidney. 24-hour ambulatory blood pressure monitoring, Bio-impedancemetry will be evaluated at T0, and T2 and the assessment of tubular oxygen consumption by MRI with BOLD method will be performed at baseline (T0) and after 12 weeks of treatment (T1). This timeline seems to be more appropriate for investigating chances in functional parameters such as blood pressure behaviour, distribution of body water and tubular oxigen consumption.

Based on health claims data published in scientific journals, the treatment extension with Dapaglifozin will be proposed to patients of both arms of the Study at the end of 24 Weeks of treatment (T2) for additional 48 Weeks (T3, T4).

ELIGIBILITY:
Inclusion Criteria:

* Albuminuria defined as urinary albumin:creatinine ratio ≥ 25 mg/g (or protein:creatinine ratio ≥ 30 mg/g) or albuminuria > 30 mg/24h
* eGFR > 25 and < 75 ml/minute 1.73m2
* BMI between 19 kg/m2 and 30 kg/m2
* Treatment with an ACE inhibitor and/or ARB at the maximum tolerated (for the individual subject) dose. The maximum tolerated dose for an individual subject may be less than the maximum labeled dose or may be zero if the medical reason is documented.
* Mean systolic and diastolic blood pressure (determined as the average of three replicates) must be < 180/90mmHg
* Pre-menopausal women of child-bearing potential 1 must have a negative pregnancy test performed before the inclusion in the study V e r s i o n 6 . 0 - P a g . 10 | 32
* Willingness to participate in the study (signed informed consent)

IN PARTICIPANTS WITH Type 2 Diabetes

* Clinical diagnosis of T2DM for at least 1 year
* Hemoglobin A1c (HbA1c) value of < 9.5%
* Patients treated only with metformin and/or repaglinide
* A diagnosis of Diabetic Nephropathy at renal biopsy made not more than 6 months before the screening visit (only for the subgroup of patients candidated to the second kidney biopsy)
* Proteinuria > 1g/24h (only for the subgroup of patients candidated to the second kidney biopsy)
* Hemoglobin A1c (HbA1c) value of > 6.5% (only for patients candidated to the second kidney biopsy) In PARTICIPANTS Without Type 2 Diabetes
* diagnosis of hypertension for at least 5 years

Exclusion Criteria:

* Type 1 Diabetes
* Hemoglobin A1c (HbA1c) value of > 9.5% during the Screening period (based on central laboratory measurement).
* The need for an adjunctive drugs on top on metformin and repaglinide
* Hemoglobin A1c (HbA1c) value of < 6.5% only for patients candidated to the second kidney biopsy
* Estimated glomerular filtration rate < 25 or > 75 ml/min/1.73m2 (according to the CKD-EPI) at screening
* Untreated urinary or genital infection at screening and follow-up
* Clear signs of volume depletion
* Symptomatic hypotension, or systolic blood pressure < 90 or non-controlled hypertension
* History of alcohol or drug abuse, anuria, dialysis, or acute kidney injury/acute renal failure in the 3 months prior to Screening Period
* Heart, liver or kidney transplant V e r s i o n 6 . 0 - P a g . 11 | 32
* Acute coronary syndrome, stroke, or transient ischemic attack within 3 months prior to informed consent
* Liver disease, defined by serum levels of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 3 x upper limit of normal (ULN) during screening
* Planned cardiac surgery or angioplasty within 3 months
* Cancer or medical history of cancer (except for basal cell carcinoma) within the last 5 years
* Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at time of screening leading to unstable body weight (e.g. surgery, aggressive diet regimen, etc.)
* SGLT2i treatment in the 10 weeks before the Screening Period
* Treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent
* Any uncontrolled endocrine disorder except T2DM
* Women who are pregnant or breastfeeding
* Pre-menopausal women of child bearing potential who are not willing to employ effective contraception according to 2007 CTFG Recommendations related to contraception and pregnancy testing in clinical trials from screening for all the duration of the study
* Patients with a known hypersensitivity to Dapagliflozin or other SGLT2- inhibitors, including hypersensitivity to excipients (e.g. lactose)
* History of pancreatitis, or pancreatic surgery, diabetic ketoacidosis
* Prior lower extremity amputation or current threat of amputation (eg, lower extremity ulcer and peripheral artery disease)
* History of severe hypoglycaemia and hypoglycaemia unawareness.
* Contraindication to MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Urinary proximal tubule cells changes in protein expression of inflammatory genes such as p16ink4a, TLR-4, phospho-p65, DKK3, Myostatin, TGFβ, SMAD 2,3 and MAPK pathways. | baseline and every 3 months up to 18 month
Urinary proximal tubule cells changes in genes such as type IV collagen fibronectin, TGF-β, TNF receptor 1, EMF cadherin production, NF-kB, MCP-1 , DKK3, myostatin and Activin A | baseline and every 3 months up to 18 month
Biopsy changes in the expression and location of senescence markers by immunohistochemistry | Baseline and after 6 month
  In the first six patients with T2DM, proteinuria > 1 g/day and biopsy proven diabetic kidney disese allocated to the treatment with dapagliflozin, we will investigate the following changes in expression and location of p16inkA, SA-beta-galactosidase, TNF receptor 1, EMF cadherin NF-kB.

SECONDARY OUTCOMES:
Changes in BOLD MRI | Baseline and after 3 month
  Changes in global and segmental renal oxygenation estimated by BOLD MRI (changes in R2* value defined as 1/T2*) at 12 and 24 weeks
Urinary markers of interstitial fibrosis | Baseline and every 3 months up to 18 month
  Changes in urinary markers of a proxy of interstitial fibrosis in patients with CKD (Mir 20)
Changes in urinary albumin excretion | Baseline and every 3 months up to 18 month
  Changes in urinary albumin excretion
Changes in eGFR | Baseline and every 3 months up to 18 month
  decrease of eGFR ml/min > 30%
Outcomes of blood presssure control | Baseline and every 6 months up to 18 month
  changes in blood pressure values and in the need of antihypertensive drugs

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genova, GE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russo E, Cappadona F, Maccio L, Di Vincenzo J, Piaggio M, Verzola D, Chirco G, Garibotto G, Esposito P, Viazzi F. Dapagliflozin Reduces Ambulatory Arterial Stiffness Index in CKD Patients with and Without Diabetes Independently of Blood Pressure Control: Results from the GLUcose Transport and Renal PROtection in Chronic Kidney Disease (GLUTREPRO) Trial. High Blood Press Cardiovasc Prev. 2026 Jan;33(1):117-126. doi: 10.1007/s40292-025-00764-3. Epub 2025 Dec 9. PMID 41366613